CLINICAL TRIAL: NCT01967043
Title: A Dose-regimen Finding Study to Evaluate Safety, Tolerability, Pharmacokinetics and Activity of Oraxol in Subjects With Advanced Malignancies
Brief Title: A Study to Evaluate Safety, Tolerability, Pharmacokinetics and Activity of Oraxol in Subjects With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kinex Pharmaceuticals Inc. (Industry)
Collaborators: Atlantic Research Group (Other)
Responsible Party: Sponsor
Organization: Athenex, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORAX-01-13-US
Record Dates: First submitted 2013-09-18; First posted 2013-10-22 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-12

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oraxol Arm 1 (Experimental): HM30181AK-US tablet administered as a single oral dose of xmg on Days x, y, and z of each cycle
  Paclitaxel administered as a fixed oral daily dose of xmg (nine xmg capsules) starting on Days x, y, and z of each cycle. Depending on the cohort, subjects will receive 2, 3, 4, or 5 consecutive days of paclitaxel per week.
  Interventions: Drug: Oraxol
- Oraxol Arm 2 (Experimental): HM30181AK-US tablet administered as a single oral dose of xmg daily with each dose of Paclitaxel
  Paclitaxel administered as a fixed oral daily dose of xmg (nine xmg capsules) starting on Days x, y, and z of each cycle. Depending on the cohort, subjects will receive 2, 3, 4, or 5 consecutive days of paclitaxel per week.
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — Oraxol (Paclitaxel + HM30181AK). Paclitaxel will be supplied as 30 mg capsules and HM30181AK-US will be supplied as 15 mg tablets.

SUMMARY:
This is a standard "3+3" Phase 1b study to determine the MTD of Oraxol (paclitaxel + HM30181 Methanesulfonate monohydrate) in subjects with advanced malignancies that may be metastatic or unresectable with measurable malignant lesion(s) per RECIST Version 1.1 criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. ≥ 18 years of age
3. Histologically or cytologically confirmed solid tumor that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
4. Measurable disease as per RECIST Version 1.1 criteria.
5. Adequate bone marrow reserve as demonstrated by

   * Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L
   * Platelet count ≥ 100 x 10⁹/L
   * Hemoglobin (Hgb) ≥ 9 g/L
6. Adequate liver function as demonstrated by

   * Total bilirubin of ≤ 1.5 mg/dL or ≤ 2.0 mg/dL for subjects with liver metastasis
   * Alanine aminotransferase (ALT)≤ 3 x upper limit of normal (ULN) or ≤ 5x ULN if liver metastasis is present
   * ALP ≤ 3 x ULN or ≤ 5 x ULN if bone metastasis is present
7. Adequate renal function as demonstrated by serum creatinine ≤ 1.5 x ULN, or 24-hr urine creatinine clearance calculation >60 mL/min
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
9. Life expectancy of at least 3 months
10. Subjects who are not currently taking prohibited medication
11. Women must be postmenopausal (> 12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or must be using effective contraception

Exclusion Criteria:

1. Have not recovered to ≤ Grade 1 toxicity from previous anticancer treatments or previous investigational agents
2. Received investigational agents within 14 days or 5 half-lives of the first study dosing day, whichever is longer.
3. Women of childbearing potential who are pregnant or breast feeding.
4. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, myocardial infarction within the last 6 months, unstable angina pectoris, cardiac arrhythmia, chronic pulmonary disease requiring oxygen, known bleeding disorders, or psychiatric illness/social situations that would limit compliance with study requirements
5. Significant or uncontrolled cardiovascular disease or bleeding disorder
6. Major surgery to the upper gastrointestinal (GI) tract, or have a history of GI disease or other medical condition that, in the opinion of the investigator may interfere with oral drug absorption
7. Subjects with a known history of allergy to paclitaxel. Subjects whose allergy was due to the IV solvent (such as Cremophor®) and not paclitaxel will be eligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) of Oraxol in subjects with advanced malignancies | one year

SECONDARY OUTCOMES:
To determine the recommended Phase 2 dose (RP2D) of Oraxol | one year six months

CONTACTS AND LOCATIONS:
Overall Officials: Min-Fun Rudolf Kwan, MD, Study Director — Kinex Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - University of Colorado Cancer Center, Aurora, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No